CLINICAL TRIAL: NCT00217724
Title: A Double-blinded Pilot Study of Glutamine for the Prevention of Paclitaxel-Induced Myalgias and Arthralgias
Brief Title: Glutamine in Preventing Myalgia and/or Arthralgia in Patients Who Are Receiving Paclitaxel For Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Only able to accrue just 18 of the 40 target & funds were limited.
Sponsor: OHSU Knight Cancer Institute (Other)
Responsible Party: Principal Investigator, Joseph Bubalo, PharmD, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: CDR0000446073; OHSU-ONC-99037-L (Other: OHSU Knight Cancer Institute); 1252 (Other: OHSU IRB)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Results first posted 2010-09-24 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Pain; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; pain
MeSH Terms: conditions — Pain | interventions — Glutamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glutamine Arm (Experimental): Beginning on day 2 of course 1 of paclitaxel administration, patients receive oral glutamine three times daily for 4 days.
  Interventions: Dietary Supplement: glutamine
- Placebo arm (Placebo Comparator): Beginning on day 2 of course 1 of paclitaxel administration, patients receive oral placebo three times daily for 4 days.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: glutamine — Given orally
  Arms: Glutamine Arm
Other: placebo — Given orally
  Arms: Placebo arm

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Nutritional supplements, such as glutamine, may prevent side effects caused by chemotherapy.

PURPOSE: This randomized clinical trial is studying glutamine to see how well it works compared to placebo in preventing myalgia and/or arthralgia in patients who are receiving paclitaxel for cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of glutamine supplementation vs placebo, in terms of prevention of paclitaxel-induced myalgia and/or arthralgia, in patients with cancer.

Secondary

* Compare the attenuation of myalgia and/or arthralgia in patients who experience myalgia and/or arthralgia treated with these regimens.

OUTLINE: This is a randomized, double-blind, crossover, pilot study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Beginning on day 2 of course 1 of paclitaxel administration, patients receive oral glutamine three times daily for 4 days.
* Arm II: Beginning on day 2 of course 1 of paclitaxel administration, patients receive oral placebo three times daily for 4 days.

Both arms crossover during course 2. In both arms, treatment continues in the absence of unacceptable toxicity.

After completion of study treatment, patients are followed for 7-10 days.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria.

* Signed informed patient consent
* Adult patients (Age > 18 years old) with a neoplastic disorder requiring paclitaxel as part of therapy, whether curative or palliative intent.
* Patients must have > 2 additional planned courses of paclitaxel.
* Patients may be out-patient or in-patient at the time of enrollment.
* Patient must have had myalgias and/or arthralgias with the most recent course(s) of paclitaxel. Paclitaxel must be being administered over 3 hours or less for each infusion.
* Patients may have chronic pain but they must be able to differentiate it from either myalgias or arthralgias and be on a stable medication regimen for pain management.
* Eastern Cooperative Group (ECOG) Performance status score < 3
* If consenting for the laboratory portion of the study the participant must have normal creatinine phosphokinase within 14 days of study entry.
* The patient, if sexually active, must be willing to agree to use an approved form of birth control.

Exclusion criteria.

* The patient has received another investigational drug within the past 30 days.
* No myalgias or arthralgias in prior paclitaxel courses.
* The patient has uncontrolled (over the last 30 days), clinically significant confounding medical conditions such as rheumatoid disease, fibromyalgia, or chronic fatigue syndrome. Also if the patient has a viral infection, cold symptoms, fever (> 38 C -degrees celsius) or influenza.
* Patients with existing neuropathies or neurologic disorders which would prevent them from accurately assessing the onset or extent of myalgias and arthralgias.
* The patient has had significant medical intervention in the last 30 days
* The patient is pregnant or lactating.
* Patients who are unable to take oral medications or with medical conditions that might inhibit their ability to absorb protein from the gastrointestinal tract.
* Patients who are unwilling to abstain from additional protein supplements of any kind other than that obtained through "normal" dietary intake.
* Patients required to take nonsteroidal anti-inflammatory agents (NSAIDS), antioxidant vitamins, and unable or unwilling to abstain from them for 1 week prior to and during glutamine/placebo therapy.
* Patients with metabolic errors or abnormalities of protein metabolism.
* Patients with a history of blood urea nitrogen level > 2 times normal with a normal serum creatinine.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 1999-07; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Bubalo, PharmD, BCPS, BCOP, Study Chair — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from oncology clinics at OHSU.
Groups:
- Oral Glutamine x 4 Days: Oral glutamine 10g powder (dissolved in 8 oz orange juice) three times daily for 4 days starting day 2 of course 1 during Paclitaxel treatment.
- Oral Placebo x 4 Days: Oral placebo 10g powder (dissolved in 8 oz orange juice) three times daily for 4 days starting day 2 of course 1 during Paclitaxel treatment.
Period: Course 1, (Glutamine/Placebo Arms)
Arm/Group | Oral Glutamine x 4 Days | Oral Placebo x 4 Days
Started | 8 | 10
Completed | 5 | 9
Not Completed | 3 | 1
Period: Course 2, (Glutamine/Placebo Crossover)
Arm/Group | Oral Glutamine x 4 Days | Oral Placebo x 4 Days
Started | 9 | 5
Completed | 8 | 5
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes those randomized to Arms 1 and 2 in both course 1 and 2.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18
Cancer Diagnosis [Number; unit: Participants] — Type of cancer diagnosis enrolled subject was receiving treatment for
  Participants
    Breast | 11
    Ovarian | 5
    Esophageal | 1
    Uterine sarcoma | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response From Glutamine Preventing Paclitaxel Induced Myalgias or Arthralgias After 2 Courses of Chemotherapy
Description: Complete Response (CR): Complete absence of myalgias or arthralgias Partial Response (PR): Myalgias and/or arthralgias occur but are attenuated in the cycle in which they receive active therapy by > 50% Stable Disease (SD): Less than 25% change in incidence, duration, or severity of myalgias/arthralgias Progressive Disease (PD): Symptoms worsen by >25% from baseline scores
Time Frame: 2 courses of chemotherapy (6 weeks)
Population: Fourteen of the 18 patients enrolled received both cycles of therapy and were thus evaluable for the primary endpoint
Measure: Number; unit: participants
Groups:
- Oral Glutamine x 4 Days: Oral glutamine 10g powder (dissolved in 8 oz orange juice) three times daily for 4 days.
- Oral Placebo x 4 Days: Oral placebo 10g powder (dissolved in 8 oz orange juice) three times daily for 4 days.
Arm/Group | Oral Glutamine x 4 Days | Oral Placebo x 4 Days
Number analyzed (Participants) | 14 | 14
participants
  Complete Response | 0 | 0
  Partial Response | 3 | 4
  Stable Disease (SD)/Progressive Disease (PD) | 11 | 10

2. Secondary Outcome: Number of Participants With Attenuation of Myalgias or Arthralgias Not Receiving Glutamine as Measured by Pain Scale Diaries on Days 1 and 3 of Courses 1 and 2
Time Frame: Duration of participation on study (up to one year)
Arm/Group | Oral Glutamine x 4 Days | Oral Placebo x 4 Days
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the life of the study (3/2002-2/2007).
Arm/Group | Oral Glutamine x 4 Days | Oral Placebo x 4 Days
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

LIMITATIONS AND CAVEATS:
We were able to only accrue 18 of the 40 patient target. This, plus confounded results and limited funds, the remaining research funds were returned to the sponsor and no evaluation of serum or dietary glutamine levels was done.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No